CLINICAL TRIAL: NCT03301233
Title: The Effect of Estradiol Valerate With and Without Oral Sildenafil on Endometrial Thickness and Pregnancy Rates in Infertile Women: A R.C.T
Brief Title: Effect Sildenafil and Estradiiol Valerate on Endometrial Thickness in Infertile Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hayam Fathy Mohammad, Assistant Professor of Obstetrics and Gynecology , Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2
Record Dates: First submitted 2017-09-24; First posted 2017-10-04 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Endometrial Thickness
MeSH Terms: interventions — Estradiol; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant
Masking Description: Ninety opaque envelopes will be numbered serially and in each envelope the corresponding letter which denotes the allocated group will be put according to randomization table. Then all envelopes will be closed and put in one box. When the first patient arrives, the first envelope will be opened and the patient will be allocated according to the letter inside.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- estradiol valerate (Active Comparator): oral estradiol valerate (Cyclo-Progynova ® 2mg, white tablets, BAYER Schering Pharma). One tablet every 12 hour from 2nd day of the cycle till the day of trigger of ovulation).
  Interventions: Drug: estradiol valerate and sildenafil
- estradiol valerate and sildenafil (Experimental): oral estradiol valerate (Cyclo-Progynova ® 2mg, white tablets, BAYER Schering Pharma), one tablet every 12 hour from 2nd day of the cycle + sildenafil (silden® 25 mg, E.I.P.I.CO.) every 8 hour from 2nd day of the cycle till the day of trigger of ovulation).
  Interventions: Drug: estradiol valerate and sildenafil

INTERVENTIONS:
Drug: estradiol valerate and sildenafil — (45 women will receive clomiphene citrate (clomid 50mg ®, Sanofi aventis) 2 tab. single dose orally from the 2nd day of the cycle for 5 days with oral estradiol valerate (Cyclo-Progynova ® 2mg, white tablets, BAYER Schering Pharma), one tablet every 12 hour from 2nd day of the cycle + sildenafil (silden® 25, E.I.P.I.CO.) every 8 hour from 2nd day of the cycle till the day of trigger of ovulation).
  Other Names: cycloprogenova and silden

SUMMARY:
The endometrium is a dynamic tissue that responds to changing hormonal signals throughout the cycle. The changes in the endometrial composition are expressed in alteration in gene expression, micro architectural morphological changes as well as in protein and hormone secretion. These factors combine together to construct the "window of implantation" a short period of time during the luteal phase in which the endometrium is receptive.

Thin endometrium is associated with a low pregnancy rate. Endometrial thickness 7 mm in the pre-ovulatory phase is widely accepted to be cut-off of thin endometrium.

for that the aim of this study is to compare the effect of sildenafil-estrogen combination to estrogen alone on endometrium thickness in infertile women. Half of the patients will receive estrogen ( estradiol valerate ) and the other half will receive combination of sildenafil-estrogen .

DETAILED DESCRIPTION:
Being a hormone dependent tissue, the endometrium proliferates in response to estrogen, which further induces the production of progesterone receptors. As a result, infertile patients who demonstrated thin endometrium, were offered estradiol (E2) remedies, in an attempt to improve endometrial proliferation. Most of the studies regarding E2 treatment in patients with thin endometrium dealt with frozen-thawed embryo transfer cycles. Moreover, while there are several routes and duration of administration of E2, including per Os, transdermal, Intramuscular and vaginal, no compelling advantage for one protocol for endometrial preparation over another, with regard to pregnancy rates, has been established.

Sildenafil acts as a type 5-specific phosphodiesterase inhibitor hence augments the vasodilatory effects of nitric oxide by preventing the degradation of cGMP. Nitric oxide (NO) relaxes vascular smooth muscle through a cGMP-mediated pathway and NO synthase isoforms have been identified in the uterus. A decade ago, Sher and Fisch studied the effect of vaginal sildenafil on the endometrial thickness of infertile patients with poor endometrial development, who underwent IVF treatment. They have demonstrated improved uterine artery blood flow and endometrial growth, with higher implantation and ongoing pregnancy rates following vaginal sildenafil administration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having ovulatory infertility.
2. Age: 20-35 years old.
3. BMI less than 30 kg/m2

Exclusion Criteria:

1. Women who have any congenital uterine anomaly (e.g., unicornuate uterus or infantile uterus) or acquired deformities of the uterine cavity that interfere with embryo implantation (as Asherman Syndrome).
2. Women who have any tubal factor that relates to infertility (e.g., tubal adhesion or previous ectopic pregnancy).
3. Women who have contraindication for estrogen treatment (e.g., history of stroke, DVT and Benign liver disease).
4. Women who have male factor for infertility (e.g., azoospermia, teratospermia).

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
endometrial line thickness | 9 days
  The thickness of the endometrium will be measured (maximum distance between each myometrial/endometrial interface through the longitudinal axis of the uterus) using two dimensional transvaginal ultrasound.

SECONDARY OUTCOMES:
positive pregnancy test | 14 days after triggering of ovulation
  Serum B-HCG
sub endometrial blood flow | 9 days
  Using two dimensional (2D) transvaginal Doppler, flow velocity wave forms will be obtained from the ascending main branch of the uterine artery on the right and left side of the cervix before it enters the uterus.

CONTACTS AND LOCATIONS:
Overall Officials: Hayam F Mohammad, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt